CLINICAL TRIAL: NCT06600971
Title: The Effect of Self Acupressure on Fatigue and Sleep Quality in Patients With Multiple Sclerosis
Brief Title: The Effect of Self Acupressure in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Gülden Atan, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS-GULDEN
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Acupressure; Fatigue; Sleep Quality
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The intervention and control groups were selected by drawing lots
Who Masked: Participant, Investigator
Masking Description: The information indicating that the patients included in the research sample were assigned to groups A and B according to the randomization table was placed in an opaque envelope. This envelope was kept by the neurology clinic secretariat. When the researcher went to the patient selected for acupressure application, he first applied a pre-test and then contacted the neurology clinic secretariat to learn which group the patient was in. In this way, the participants were blinded in terms of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure (Experimental): The patients in the experimental group received acupressure application for a total of 8 sessions, 2 sessions per week. The first application was performed in a room in the polyclinic by a researcher with an acupressure application certificate. Immediately after the preparation phase, the researcher applied acupressure with the thumb in a certain order (Ht7-Ht7 and St36-St36) on each point to be pressed, in accordance with the acupressure application protocol, for a duration of 2 minutes. Verbal communication was maintained during the procedure to ensure the patient's relaxation. After the first application, the application was taught to the patient. In addition, the researcher established a WhatsApp group for regular follow-up of the patients in the experimental group, and the video recording of the acupressure was sent to the patients and they were asked to watch it.
  Interventions: Other: acupressure application
- Control (No Intervention): During the study, it was explained to the control group that their fatigue and sleep quality levels would be monitored for four weeks without any intervention (other than routine treatment given by the physician). Patients in this group were asked to fill out the Fatigue Severity Scale and the Richard-Campbell Sleep Scale at the beginning and again in the 4th week.

INTERVENTIONS:
Other: acupressure application — The patients in the experimental group received acupressure application for a total of 8 sessions, 2 sessions per week.
  Arms: acupressure

SUMMARY:
Patients with MS use non-pharmacological methods as well as pharmacological methods in the treatment of their symptoms. Acupuncture, acupressure, aquatherapy, reflexology and aromatherapy are also complementary and integrated methods frequently used in patients with MS. Integrated methods, which have an important place in independent nursing practices, have been preferred in nursing practices in recent years due to their safety, ease of application and minimal side effects. In addition, acupressure application is included in the Nursing Interventions Classification, and is a method that increases the independent functions of the nurse and improves patient-nurse interaction.

DETAILED DESCRIPTION:
In addition to pharmacological methods, patients with MS also use non-pharmacological methods in the treatment of the symptoms they experience. Acupuncture, acupressure, aquatherapy, reflexology and aromatherapy are also complementary and integrated methods frequently used in MS. Integrated methods, which have an important place in independent nursing practices, have been preferred in nursing practices in recent years due to their safety, ease of application and minimal side effects. In addition, acupressure application is included in the Nursing Interventions Classification (NIC), and is a method that increases the independent functions of the nurse and improves patient-nurse interaction. In addition, it is reported that acupressure, which is used in symptom control, should be used in care plans by nurses because it is one of the integrated methods. Acupressure, one of the integrated treatment methods used for many years, can be applied to increase sleep quality and reduce fatigue levels. Acupressure is a massage technique based on the principle of applying pressure to specific points on the body using hands, fingers and stimulator tools. It has been determined that acupressure, which is reported to be applied safely by nurses in the literature, is effective in controlling fatigue, pain, sleep quality, depression, anxiety, quality of life and stress levels of patients with MS. Therefore, nurses should be able to apply integrated methods in the management of symptoms experienced by patients with MS in cooperation with other members of the healthcare team and inform patients about these methods. It is believed that the results of the study to be conducted on this subject will contribute to nursing interventions in the symptom management of MS.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* Those who can read and write,
* Those who can speak Turkish,
* Patients diagnosed with multiple sclerosis,
* Patients who do not have a neurological disease other than MS,
* Those who volunteer to participate in our study,
* Patients who are conscious and do not have a psychiatric health problem

Exclusion Criteria:

* • Patients with nerve, soft tissue, vascular disease infections in their extremities, who have undergone surgery,

  * Patients with bleeding problems, pacemaker or heart failure and a diagnosed condition, mass and flattening in the neck,
  * Patients with a diagnosis other than MS (such as subarachnoid hemorrhage, aneurysm, dementia, a psychiatric disease),
  * Patients who have had a hemorrhagic stroke,
  * Patients with malignancy,
  * Patients with vision and hearing problems,
  * Patients who do not volunteer to participate in our study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 4 weeks
  The scale is a Likert type with 9 questions, and each question is rated from 1 (strongly disagree) to 7 (strongly agree). The total score varies between 9-63, with total scores of 27 and above indicating fatigue.
Richard-Campbell Sleep Scale | 4 weeks
  The scale consists of 6 items. The items measure the depth of night sleep, the time it takes to fall asleep, the frequency of waking up, the time it takes to stay awake when you wake up, the quality of sleep, and the noise level in the environment. A score of "0-25" indicates "very bad sleep", and a score of "76-100" indicates "very good sleep". While the total score of the scale is calculated, the scores from the 5 items are added up, and the 6th item is not included in the total score evaluation. The minimum score from the scale is 0 and the maximum score is 100. An increase in the score from the scale indicates an increase in sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Gülden Atan, PHD, Principal Investigator — Faculty of health science, Yuzuncu Yıl University , Van, TURKEY.
Locations (1):
- Yuzuncu Yıl University , Faculty of health science, Van, Turkey (Türkiye)